CLINICAL TRIAL: NCT04866160
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Rising Oral Doses of BI 1291583 qd Versus Placebo in Healthy Male and Female Subjects for 4 Weeks (Single-blind, Partially Randomised, Placebo-controlled Parallel Group Design)
Brief Title: A Trial in Healthy Men and Women to Find Out How Well Different Doses of BI 1291583 Are Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1397-0011; 2020-006070-74 (EudraCT Number)
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BI 1291583 low dose (Experimental)
  Interventions: Drug: BI 1291583
- BI 1291583 high dose (Experimental)
  Interventions: Drug: BI 1291583
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1291583 — BI 1291583
  Other Names: Verducatib
  Arms: BI 1291583 high dose; BI 1291583 low dose
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics (PK) of BI 1291583 in healthy male and female subjects following administration of multiple rising doses over 4 weeks and to explore the pharmacokinetics (PK) and pharmacodynamics (PD) of BI 1291583 after multiple dosing and assess the PK/PD relationship.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Male, or female (of non-childbearing potential) subjects

For 'female of non-childbearing potential' at least one of the following criteria must be fulfilled:

* Permanently sterile (permanent sterilisation methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy)
* Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR, or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Number (N) of subjects with drug-related AEs | up to 77 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over a uniform dosing interval τ after administration of the first dose (AUCτ,1) | up to 24 hours
Maximum measured concentration of the analyte in plasma after administration of the first dose (Cmax,1) | up to 24 hours
Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) | at day 28
Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmax,ss) | at day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Fraunhofer ITEM, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com